CLINICAL TRIAL: NCT05324202
Title: New Imaging Procedures and Therapeutic Approach in Basal Cell Carcinoma
Brief Title: New Imaging Procedures and Therapeutic Approach in Basal Cell Carcinoma Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Stephanie Geisler (Other)
Responsible Party: Sponsor-Investigator, Dr. Stephanie Geisler, Investigator, Resident in Dermatology, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ndyag_BCC_1
Record Dates: First submitted 2021-10-05; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nd:YAG treatment arm (Other)
  Interventions: Device: Cynosure Cynergy Nd:YAG Laser 1064nm

INTERVENTIONS:
Device: Cynosure Cynergy Nd:YAG Laser 1064nm — The Nd:YAG Laser 1064nm is intended to be used as a treatment option in individuals suffering from low-risk basal cell carcinoma(s).

SUMMARY:
The aim of this study is to show that the Nd:YAG laser could be a promising alternative treatment option in the management of low-risk basal cell carcinomas with similar high efficacy rates to surgery, and low recurrence rates evaluated over a time period of one year. Reflectance confocal microscopy, optical coherence tomography and clinical examination are used prior to confirm the clinical diagnosis of the basal cell carcinoma and for premargination of the tumor. The optical coherence tomography will also be used post treatment to confirm clearance of the basal cell carcinoma and to monitor treatment response.

ELIGIBILITY:
Inclusion Criteria:

Patients with one or more basal cell carcinoma(s) on head, trunk or extremities

* Diagnosed clinically, with a dermatoscope and through noninvasive imaging methods such as reflectance confocal microscopy and optical coherence tomography
* H zone <6mm, M zone <10mm, L zone <20mm
* Tumor thickness <2mm
* Clearly visible margins

Exclusion Criteria:

* Pregnancy
* <18 years of age
* Current or history of immunosuppression
* Prior-treatment of the basal cell carcinoma/ recurrent basal cell carcinomas
* History of radiation in the area of basal cell carcinoma appearance

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy of Nd:YAG Laser 1064-nm for low risk basal cell carcinomas | 8 weeks after the treatment
  Clearance rate of basal cell carcinomas after 1-3 Nd:YAG laser treatments evaluated by clinical inspectation, dermatosopy and optical coherence tomography.
Recurrence Rate after Nd:YAG Laser treatment | 12 months
  To assess the recurrence rate after a long-term follow-up of 6 and 12 months

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 6 and 12 months after treatment
  To assess treatment tolerability of the Nd:YAG Laser 1064-nm (e.g. pain according to a Numerical rating scale, scarring, wound healing, secondary infection rate)
Cosmetic outcome after laser treatment | 6 and 12 months after treatment
  This will be assess according to an assessment scale including following parameters:
  * Pigmentation: hyperpigmentation, hypopigmentation, normal
  * Vascularity: pink, red, purple, normal
  * Pliability: firm, contracture, supple, yielding, ropes, normal
  * Scarring: yes, no
  * Overall opinion: Rating on a scale from 1-5 (school note system) Separate evaluation of observer and patient.